CLINICAL TRIAL: NCT02571452
Title: Telephone-Facilitated Insomnia Treatment in Primary Care for OEF/OIF/OND Veterans
Brief Title: Brief Behavioral Insomnia Treatment Study
Acronym: BBTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D1539-I
Record Dates: First submitted 2015-10-02; First posted 2015-10-08 (Estimated); Results first posted 2020-01-22 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-01

CONDITIONS: Insomnia Disorder
Keywords: Veteran; Insomnia; Primary Healthcare
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Autogenic Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brief Behavioral Treatment for Insomnia (Experimental): Participants will receive 4 weeks of Brief Behavioral Treatment for Insomnia (BBTI). BBTI consists of two in-person sessions, with the two other sessions conducted via telephone. BBTI emphasizes behavioral elements of insomnia treatment. Treatment begins with sleep education and discussion of the biological rhythms that influence sleep cycles. Next, a series of interventions are employed that are derived from sleep restriction and stimulus control techniques.
  Interventions: Behavioral: Brief Behavioral Treatment for Insomnia
- Progressive Muscle Relaxation (Active Comparator): Participants will receive 4 weeks of progressive muscle relaxation training (PMRT). PMRT consists of two in-person and two phone sessions. Treatment begins with training on muscle tensing and relaxing, and advances to progressively more efficient tensing-relaxing and passive relaxation exercises. Sessions are employed that teach techniques and problem-solve barriers to the use of PMRT.
  Interventions: Behavioral: Progressive Muscle Relaxation

INTERVENTIONS:
Behavioral: Brief Behavioral Treatment for Insomnia — Participants will receive 4 weeks of Brief Behavioral Treatment for Insomnia (BBTI). BBTI consists of two in-person sessions, with the two other sessions conducted via telephone. BBTI emphasizes behavioral elements of insomnia treatment. Treatment begins with sleep education and discussion of the biological rhythms that influence sleep cycles. Next, a series of interventions are employed that are derived from sleep restriction and stimulus control techniques.
  Arms: Brief Behavioral Treatment for Insomnia
Behavioral: Progressive Muscle Relaxation — Participants will receive 4 weeks of progressive muscle relaxation training (PMRT). PMRT consists of two in-person and two phone sessions. Treatment begins with training on muscle tensing and relaxing, and advances to progressively more efficient tensing-relaxing and passive relaxation exercises. Sessions are employed that teach techniques and problem-solve barriers to the use of PMRT.
  Arms: Progressive Muscle Relaxation

SUMMARY:
The purpose of this study is to determine whether a brief, behavioral treatment for insomnia is effective in addressing social and occupational functioning and overall health among Veterans with insomnia disorder.

DETAILED DESCRIPTION:
This study is a randomized, controlled trial of a telephone-based, brief insomnia treatment in primary care in order to accomplish the goal of improving psychosocial functioning in Veterans who meet criteria for Insomnia Disorder. The primary outcome for the trial will be psychosocial functioning, with insomnia severity serving as the secondary outcome. Additional goals include evaluating durability of treatment gains and obtaining feedback from participants about the utility and feasibility of the proposed insomnia treatment.

ELIGIBILITY:
Inclusion Criteria:

* Veterans between the ages of 18-75 years.
* Meet DSM-5 Criteria for Insomnia Disorder.
* Able attend in-person appointments at the San Francisco VA Medical Center
* The investigators will not exclude individuals who are taking insomnia or antidepressant medications, provided they have been stable on these medications for at least one month and still meet criteria for Insomnia Disorder as described above.

  * Specifically, individuals receiving benzodiazepine or benzodiazepine receptor agonists, anticonvulsants, atypical antipsychotic medication, or non-SSRI antidepressant medications such as trazodone will not be excluded provided they meet the criteria described above.
* The investigators will not exclude Veterans receiving any type of psychotherapy, provided they have received this treatment for at least three months and do not plan to discontinue this treatment during the BBTI trial.

  * However, individual who need to start a new type of psychotherapy during the course of the treatment will be excluded, or they will need to wait three months in order to enroll in the trial.
* The investigators will not exclude individuals with TBI.
* The investigators will not exclude individuals with chronic pain.
* The investigators will not exclude individuals based on any other mental health condition, including posttraumatic stress disorder and depression.

Exclusion Criteria:

* Conditions that may be associated with comorbid insomnia, including a lifetime history of any psychiatric disorder with psychotic features or bipolar disorder, and alcohol or drug dependence within the past year.
* Individuals who meet criteria for alcohol or drug abuse will be asked to reduce alcohol to recommended limits during the course of the study and/or refrain from drug use in order to be included.
* Veterans with suicidal or homicidal ideation.
* Veterans who are pregnant, due to the biological impact of pregnancy on sleep.
* Veterans who work night or rotating shifts.
* Veterans with untreated moderate to severe sleep apnea (those receiving treatment will not be excluded from the study).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2016-01-06 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shira Maguen, PhD, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA
Locations (1):
- San Francisco VA Medical Center, San Francisco, CA, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ranney RM, Gloria R, Metzler TJ, Huggins J, Neylan TC, Maguen S. Brief behavioral treatment for insomnia decreases trauma-related nightmare frequency in veterans. J Clin Sleep Med. 2022 Jul 1;18(7):1831-1839. doi: 10.5664/jcsm.10002. PMID 35393934
- [Derived] Maguen S, Gloria R, Huggins J, Goldstein LA, Kanady JC, Straus LD, Metzler TJ, Lujan C, Neylan TC. Brief behavioral treatment for insomnia improves psychosocial functioning in veterans: results from a randomized controlled trial. Sleep. 2021 Mar 12;44(3):zsaa205. doi: 10.1093/sleep/zsaa205. PMID 33022048

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 1/6/16 to 8/9/18 through local advertisements, referrals from other research studies or VA clinicians and direct mailings to veterans that had established care at the San Francisco VA (SFVA) or that lived within a 40-mile radius of the SFVA.
Pre-assignment Details: A total of 157 people provided consent for screening, 119 completed screening and 93 were eligible, enrolled and randomized to treatment. Of the 93, two were withdrawn during treatment or 6-month follow-up due to no longer meeting eligibility and two were pilot subjects that didn't meet inclusion criteria and weren't included in data analysis.
Groups:
- Progressive Muscle Relaxation Training: Participants will receive 4 weeks of progressive muscle relaxation training (PMRT). PMRT consists of two in-person and two phone sessions. Treatment begins with training on muscle tensing and relaxing, and advances to progressively more efficient tensing-relaxing and passive relaxation exercises. Sessions are employed that teach techniques and problem-solve barriers to the use of PMRT.
  Progressive Muscle Relaxation: Participants will receive 4 weeks of progressive muscle relaxation training (PMRT). PMRT consists of two in-person and two phone sessions. Treatment begins with training on muscle tensing and relaxing, and advances to progressively more efficient tensing-relaxing and passive relaxation exercises. Sessions are employed that teach techniques and problem-solve barriers to the use of PMRT.
Period: Overall Study Treatment
Arm/Group | Brief Behavioral Treatment for Insomnia | Progressive Muscle Relaxation Training
Started (Randomized to Treatment Arm) | 47 | 46
Completed (Completed Treatment) | 47 | 45
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1
Period: Overall Study 6-Month Follow-up
Arm/Group | Brief Behavioral Treatment for Insomnia | Progressive Muscle Relaxation Training
Started (Scheduled for 6-Month Follow-up Assessment) | 47 | 0 (Participants in the PMRT arm were not invited to complete 6-Month Follow-up.)
Completed | 42 | 0
Not Completed | 5 | 0
Not completed — Lost to Follow-up | 4 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: One participant in each group was a pilot participant that didn't meet all inclusion criteria. Therefore, these two individuals were not included in data analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Brief Behavioral Treatment for Insomnia | Progressive Muscle Relaxation Training | Total
Number analyzed (Participants) | 47 | 46 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One participant in each group was a pilot participant that didn't meet all inclusion criteria. Therefore, these two individuals were not included in data analysis.
  years
    number analyzed (Participants) | 46 | 45 | 91
    (all) | 48.87 (15.66) | 49.80 (15.46) | 49.32 (15.48)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One participant in each group was a pilot participant that didn't meet all inclusion criteria. These two individuals were not included in data analysis. Additionally, these categories exclude 1 transgender participant in the PMRT group, so the numbers below only reflects the individuals that identified as male or female.
  Participants
    number analyzed (Participants) | 46 | 44 | 90
    Female | 9 | 8 | 17
    Male | 37 | 36 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: One participant in each group was a pilot participant that didn't meet all inclusion criteria. Therefore, these two individuals were not included in data analysis.
  Participants
    number analyzed (Participants) | 46 | 45 | 91
    Hispanic or Latino | 6 | 5 | 11
    Not Hispanic or Latino | 39 | 38 | 77
    Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: One participant in each group was a pilot participant that didn't meet all inclusion criteria. Therefore, these two individuals were not included in data analysis.
  Participants
    number analyzed (Participants) | 46 | 45 | 91
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 10 | 7 | 17
    Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
    Black or African American | 8 | 4 | 12
    White | 22 | 24 | 46
    More than one race | 3 | 5 | 8
    Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Number; unit: participants] — Population: One participant in each group was a pilot participant that didn't meet all inclusion criteria. Therefore, these two individuals were not included in data analysis.
  participants
    United States: number analyzed (Participants) | 46 | 45 | 91
    United States | 46 | 45 | 91

OUTCOME MEASURES:

1. Primary Outcome: Work and Social Adjustment Scale (WSAS)
Description: The WSAS assesses functioning at work, home, management, social leisure activities, private leisure activities, and relationships with others. Scores range from 0-40, with higher scores meaning greater impairment. The measure was administered at Baseline (week 0), Mid-treatment (week 3) & Post-treatment (week 5).
Time Frame: Change from Mid-treatment to Post-treatment (week 3 to week 5), with Baseline as a covariate
Population: An intent-to-treat analysis was conducted on all participants that started treatment (91), not including the two pilot participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brief Behavioral Treatment for Insomnia | Progressive Muscle Relaxation
Number analyzed (Participants) | 46 | 45
score on a scale
  Baseline | 20.1 (9.6) | 19.7 (8.9)
  Mid-Treatment: number analyzed (Participants) | 46 | 44
  Mid-Treatment | 14.1 (9.1) | 15.8 (9.5)
  Post-Treatment: number analyzed (Participants) | 46 | 44
  Post-Treatment | 10.8 (9.3) | 14.1 (10.0)
Statistical Analysis 1: Comparison: Brief Behavioral Treatment for Insomnia vs Progressive Muscle Relaxation; Test type: Superiority; p = .021, Mixed Models Analysis — The threshold for statistical significance was p=.05; Mean Difference (Net) = -3.60, 95% CI 2-sided [-6.65 to -0.55], Standard Error of Mean 1.53

2. Primary Outcome: Work and Social Adjustment Scale (WSAS)
Description: The WSAS assesses functioning at work, home, management, social leisure activities, private leisure activities, and relationships with others. Scores range from 0-40, with higher scores meaning greater impairment. The WSAS was administered at Follow-up (6 months Post-treatment) for participants receiving the experimental treatment only.
Time Frame: Change from Post-treatment to Follow-up (after 6 months)--for treatment arm only
Population: An intent-to-treat analysis was conducted on the 46 participants that completed BBTI treatment. Participants in the PMRT group did not complete the 6-month follow-up assessment and were not included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brief Behavioral Treatment for Insomnia | Progressive Muscle Relaxation
Number analyzed (Participants) | 46 | 0
score on a scale
  Post-Treatment | 10.8 (9.3) |
  6-month follow-up: number analyzed (Participants) | 42 | 0
  6-month follow-up | 11.2 (10.3) |
Statistical Analysis 1: Comparison: Brief Behavioral Treatment for Insomnia; Test type: Superiority; p = .568, Mixed Models Analysis — The threshold for statistical significance was p=.05; Mean Difference (Net) = 0.52, 95% CI 2-sided [-1.26 to 2.30], Standard Error of Mean 0.57

3. Secondary Outcome: Insomnia Severity (ISI)
Description: The ISI is a specific index of perceived insomnia severity. Areas assessed include problems with sleep onset, sleep maintenance, and early morning awakening; dissatisfaction with sleep; interference with daily functioning; impact on quality of life; and worry about sleep problems. Scores range from 0-28, with higher scores meaning greater impairment. The measure was administered at Baseline (week 0), Mid-treatment (week 3) & Post-treatment (week 5).
Time Frame: Change from Mid-treatment to Post-treatment (week 3 to week 5), with Baseline as a covariate
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brief Behavioral Treatment for Insomnia | Progressive Muscle Relaxation
Number analyzed (Participants) | 46 | 45
score on a scale
  Baseline | 17.1 (3.6) | 17.4 (4.0)
  Mid-Treatment: number analyzed (Participants) | 46 | 44
  Mid-Treatment | 10.4 (4.6) | 14.2 (4.3)
  Post-Treatment: number analyzed (Participants) | 46 | 44
  Post-Treatment | 8.1 (5.4) | 12.4 (5.4)
Statistical Analysis 1: Comparison: Brief Behavioral Treatment for Insomnia vs Progressive Muscle Relaxation; Test type: Superiority; p < .001, Mixed Models Analysis — The threshold for statistical significance was p=.05; Mean Difference (Net) = -4.10, 95% CI 2-sided [-5.87 to -2.33], Standard Error of Mean 0.89

4. Secondary Outcome: Insomnia Severity (ISI)
Description: Insomnia Severity Index (ISI) is a specific index of perceived insomnia severity. Areas assessed include problems with sleep onset, sleep maintenance, and early morning awakening; dissatisfaction with sleep; interference with daily functioning; impact on quality of life; and worry about sleep problems. Scores range from 0-28, with higher scores meaning greater impairment. The ISI was administered at Follow-up (6 months Post-treatment) for participants receiving the experimental treatment only.
Time Frame: Change from Post-treatment to Follow-up (after 6 months)--for treatment arm only
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brief Behavioral Treatment for Insomnia | Progressive Muscle Relaxation
Number analyzed (Participants) | 46 | 0
score on a scale
  Post-Treatment | 8.1 (5.4) |
  6-month follow-up: number analyzed (Participants) | 42 | 0
  6-month follow-up | 7.5 (5.7) |
Statistical Analysis 1: Comparison: Brief Behavioral Treatment for Insomnia; Test type: Superiority; p = .173, Mixed Models Analysis — The threshold for statistical significance was p=.05; Mean Difference (Net) = -0.66, 95% CI 2-sided [-1.61 to 0.29], Standard Error of Mean 0.49

ADVERSE EVENTS:
Time Frame: Adverse events were collected beginning from participant screening to the last study visit. For the PMRT group, this was from screening to Post-treatment visits (approximately 7 weeks).For the BBTI group, this was from screening to Follow-up visits (approximately 8 months).
Arm/Group | Brief Behavioral Treatment for Insomnia | Progressive Muscle Relaxation Training
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/46
Other Adverse Events (participants affected / at risk) | 0/47 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-02): https://cdn.clinicaltrials.gov/large-docs/52/NCT02571452/Prot_SAP_000.pdf